CLINICAL TRIAL: NCT02380677
Title: Phase 1/2a Dose-Escalation Study of CRLX301 in Patients With Advanced Solid Tumor Malignancies
Brief Title: Phase 1/2a Dose-Escalation Study of CRLX301 in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company decision
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRLX301-101
Record Dates: First submitted 2015-02-19; First posted 2015-03-05 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Advanced Solid Tumor Malignancy

STUDY DESIGN:
Intervention Model Description: Phase 1 dose escalation study followed by phase 2a expansion cohort
Oversight: Data Monitoring Committee: No

ARMS (12):
- Schedule 1 Cohort 1 (Experimental): CRLX301 7.5 mg/m2 IV given every 3 weeks
  Interventions: Drug: CRLX301
- Schedule 1 Cohort 2 (Experimental): CRLX301 15 mg/m2 IV given every 3 weeks
  Interventions: Drug: CRLX301
- Schedule 1 Cohort 3 (Experimental): CRLX301 30 mg/m2 IV given every 3 weeks
  Interventions: Drug: CRLX301
- Schedule 1 Cohort 4 (Experimental): CRLX301 60 mg/m2 IV given every 3 weeks
  Interventions: Drug: CRLX301
- Schedule 1 Cohort 5 (Experimental): CRLX301 75 mg/m2 IV given every 3 weeks
  Interventions: Drug: CRLX301
- Schedule 1 Cohort 6 (Experimental): CRLX301 90 mg/m2 IV given every 3 weeks
  Interventions: Drug: CRLX301
- Schedule 2 Cohort 1 (Experimental): CRLX301 25 mg/m2 IV given weekly
  Interventions: Drug: CRLX301
- Schedule 2 Cohort 2 (Experimental): CRLX301 35 mg/m2 IV given weekly
  Interventions: Drug: CRLX301
- Schedule 2 Cohort 3 (Experimental): CRLX301 45 mg/m2 IV given weekly
  Interventions: Drug: CRLX301
- Schedule 2 Cohort 4 (Experimental): CRLX301 54 mg/m2 IV given weekly
  Interventions: Drug: CRLX301
- Schedule 2 Cohort 5 (Experimental): CRLX301 54 mg/m2 given weekly for 3 weeks with 1 week off
  Interventions: Drug: CRLX301
- Phase 2a expansion cohort (Experimental): CRLX301 75mg/m2 IV given every 3 weeks
  Interventions: Drug: CRLX301

INTERVENTIONS:
Drug: CRLX301

SUMMARY:
A Phase 1/2a, open-label, dose-escalation study with enrollment in Phase 1 to continue until determination of the Maximum Tolerated Dose (MTD) /Recommended Phase 2a Dose (RP2D), and then enrollment into Phase 2a expansion cohorts will be initiated.

DETAILED DESCRIPTION:
Phase 1 is an open-label, dose-escalation protocol. It is anticipated that up to 36 patients will be enrolled in Phase 1. All patients will be assigned to treatment with CRLX301 as the single agent.

For the first 2 cohorts a 1+5 study design will be utilized. A single patient will be enrolled sequentially into cohort 1 and cohort 2. If either patient in cohort 1 or 2 experiences a dose limiting toxicity (DLT) during Cycle 1, then the cohort will be expanded to enroll additional patients up to a total of 6.

As of cohort 3 and for all subsequent cohorts, a 3+3 dose escalation schema will be utilized.

MTD/RP2D will be determined at the dose level when <2 of 6 patients experience a DLT in a cohort.

The Phase 2a part of the study will be an open-label expansion cohort study. An additional 24 patients with advanced, histologically confirmed solid tumor malignancies will be enrolled. All patients will be assigned to treatment at the MTD/RP2D with CRLX301 as the single agent.

All patients will be followed for safety, tumor response, and progression free survival (PFS) all per RECIST version 1.1 guidelines. Patients will remain on study treatment until they experience progression of disease, unacceptable toxicity, or other specified reason for discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age
2. Diagnosis of histologically or cytologically confirmed, advanced solid tumor malignancy that is refractory to or not a candidate for standard therapy
3. ECOG 0 or 1
4. Life expectancy >12 weeks
5. Fertile males or females of childbearing potential agree to use adequate contraception prior to study entry
6. Negative urine pregnancy test

Exclusion Criteria:

1. Uncontrolled grade 2 or greater toxicity except alopecia
2. Prolongation of QT/QTc interval
3. Women who are pregnant or nursing
4. Any known HIV infection or AIDS or any concurrent infection requiring IV antibiotics
5. Any chronic or concurrent acute liver disease, including viral hepatitis
6. Primary brain malignant tumors
7. Known metastases to the brain
8. Uncontrolled hypertension
9. Concurrent participation in any other investigational study
10. Concurrent treatment with anticoagulation medication, unless approved by Sponsor
11. History of stroke, deep venous thrombosis (DVT), or transient ischemic attack (TIA)
12. History of other cancer type, except for cutaneous basal cell or squamous cell carcinoma, or cervical or prostate cancer in situ, within the last 2 years prior to C1D1
13. Uncontrolled concurrent disease or illness
14. History of severe hypersensitivity reaction to taxanes
15. Peripheral neuropathy exclusions
16. Other condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or that may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-04; Primary Completion 2017-10-04 (Actual); Study Completion 2017-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Dees, MD, Principal Investigator — University of North Carolina
Locations (3):
- United States (3):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson, Houston, Texas

REFERENCES:
- [Derived] Piha-Paul SA, Thein KZ, De Souza P, Kefford R, Gangadhar T, Smith C, Schuster S, Zamboni WC, Dees CE, Markman B. First-in-human, phase I/IIa study of CRLX301, a nanoparticle drug conjugate containing docetaxel, in patients with advanced or metastatic solid malignancies. Invest New Drugs. 2021 Aug;39(4):1047-1056. doi: 10.1007/s10637-021-01081-x. Epub 2021 Feb 16. PMID 33594602

RESULTS

PARTICIPANT FLOW:
Groups:
- Schedule 1 Cohort 1: CRLX301 7.5 mg/m2 IV given every 3 weeks
  CRLX301
- Schedule 1 Cohort 2: CRLX301 15 mg/m2 IV given every 3 weeks
  CRLX301
- Schedule 1 Cohort 3: CRLX301 30 mg/m2 IV given every 3 weeks
  CRLX301
- Schedule 1 Cohort 5: CRLX301 60 mg/m2 IV given every 3 weeks
  CRLX301
- Schedule 1 Cohort 6: CRLX301 75 mg/m2 IV given every 3 weeks
  CRLX301
- Schedule 1 Cohort 7: CRLX301 90 mg/m2 IV given every 3 weeks
  CRLX301
- Schedule 2 Cohort 1: CRLX301 25 mg/m2 IV given weekly
  CRLX301
- Schedule 2 Cohort 2: CRLX301 35 mg/m2 IV given weekly
  CRLX301
- Schedule 2 Cohort 3: CRLX301 45 mg/m2 IV given weekly
  CRLX301
- Schedule 2 Cohort 4: CRLX301 54 mg/m2 IV given weekly
  CRLX301
- Schedule 2 Cohort 5: CRLX301 54 mg/m2 given weekly for 3 weeks with 1 week off
  CRLX301
- Phase 2a Expansion Cohort: CRLX301 75mg/m2 IV given every 3 weeks
  CRLX301
Period: Overall Study
Arm/Group | Schedule 1 Cohort 1 | Schedule 1 Cohort 2 | Schedule 1 Cohort 3 | Schedule 1 Cohort 5 | Schedule 1 Cohort 6 | Schedule 1 Cohort 7 | Schedule 2 Cohort 1 | Schedule 2 Cohort 2 | Schedule 2 Cohort 3 | Schedule 2 Cohort 4 | Schedule 2 Cohort 5 | Phase 2a Expansion Cohort
Started | 1 | 1 | 3 | 3 | 6 | 6 | 3 | 4 | 4 | 2 | 4 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 3 | 3 | 6 | 6 | 3 | 4 | 4 | 2 | 4 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 4 | 2 | 2 | 2 | 1 | 2 | 1
Not completed — Physician Decision | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 2 | 0 | 4 | 1 | 1 | 2 | 2 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Not completed — Other | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Schedule 1 Cohort 1 | Schedule 1 Cohort 2 | Schedule 1 Cohort 3 | Schedule 1 Cohort 5 | Schedule 1 Cohort 6 | Schedule 1 Cohort 7 | Schedule 2 Cohort 1 | Schedule 2 Cohort 2 | Schedule 2 Cohort 3 | Schedule 2 Cohort 4 | Schedule 2 Cohort 5 | Phase 2a Expansion Cohort | Total
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 6 | 6 | 3 | 4 | 4 | 2 | 4 | 5 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (NA) — Only 1 participant | 43 (NA) — Only 1 participant | 59 (19) | 67.3 (1.53) | 63.8 (9.79) | 60.2 (11.62) | 65 (2.65) | 56 (11.52) | 54 (12.25) | 72.5 (2.12) | 60.3 (3.1) | 66.8 (4.15) | 61.8 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 1 | 2 | 4 | 3 | 1 | 2 | 0 | 1 | 0 | 16
  Male | 1 | 1 | 1 | 2 | 4 | 2 | 0 | 3 | 2 | 2 | 3 | 5 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 4
  Not Hispanic or Latino | 1 | 1 | 2 | 3 | 6 | 6 | 3 | 4 | 3 | 2 | 4 | 3 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3
  White | 1 | 1 | 3 | 3 | 6 | 4 | 3 | 3 | 3 | 1 | 4 | 5 | 37
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Primary Site of Disease at Study Entry [Count of Participants; unit: Participants]
  Bladder | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Bone | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Breast | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Hepatic/liver | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Lung | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  Lymph nodes | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Pancreas | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Pleura | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Skin | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Prostate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 5
  Other (not specified) | 0 | 1 | 3 | 0 | 3 | 1 | 2 | 3 | 1 | 0 | 3 | 1 | 18
  Abdomen/peritoneum | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Baseline ECOG Status [Count of Participants; unit: Participants] — Patients were assessed by systemic assessment using the ECOG performance scale. All patients had to be 0 or 1 for inclusion in the study. ECOG performance score of 0 = Fully active, able to carry on all pre-disease performance without restriction. ECOG performance score of 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work, etc.
  Participants
    ECOG PS Score 0 | 0 | 0 | 2 | 1 | 4 | 3 | 1 | 1 | 3 | 0 | 1 | 1 | 17
    ECOG PS Score 1 | 1 | 1 | 1 | 2 | 2 | 3 | 2 | 3 | 1 | 2 | 3 | 4 | 25
Baseline BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 30.255 (NA) — Only 1 participant | 19.63 (NA) — Only 1 participant | 28.023 (1.2871) | 26.917 (7.6956) | 26.779 (4.8762) | 27.422 (2.7810) | 33.869 (5.5301) | 25.173 (5.7256) | 24.340 (3.1519) | 28.142 (3.4551) | 26.758 (4.9670) | 29.118 (8.0521) | 27.783 (3.2805)

OUTCOME MEASURES:

1. Primary Outcome: Number of Phase 1 Participants With Treatment Emergent Adverse Events and Dose Limiting Toxicities
Description: Determination of MTD is dependent upon number of dose limiting toxicities and significant adverse events observed.
Time Frame: 13 to 19 months
Population: The phase 1 safety population were analyzed for dose limiting toxicities and treatment emergent adverse events. Treatment totals include all patients that received the specific dose at any point during the study.
Measure: Number; unit: Patients with event
Arm/Group | Schedule 1 Cohort 1 | Schedule 1 Cohort 2 | Schedule 1 Cohort 3 | Schedule 1 Cohort 5 | Schedule 1 Cohort 6 | Schedule 1 Cohort 7 | Schedule 2 Cohort 1 | Schedule 2 Cohort 2 | Schedule 2 Cohort 3 | Schedule 2 Cohort 4 | Schedule 2 Cohort 5
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 6 | 6 | 3 | 4 | 4 | 2 | 4
Patients with event
  At least one TEAE | 1 | 1 | 3 | 3 | 6 | 6 | 3 | 4 | 4 | 2 | 4
  At least one Serious TEAE | 0 | 1 | 3 | 3 | 1 | 3 | 1 | 2 | 1 | 1 | 0
  At least one DLT | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  At least one severe TEAE | 0 | 1 | 3 | 3 | 4 | 6 | 0 | 2 | 2 | 2 | 4
  At least one related TEAE | 1 | 1 | 2 | 3 | 6 | 6 | 3 | 3 | 4 | 2 | 4
  At least one TEAE leading to discontinuation | 0 | 0 | 0 | 2 | 1 | 4 | 2 | 1 | 2 | 1 | 0

2. Primary Outcome: Number of Phase 2a Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Safety variables will include AEs, SAEs, Severe AEs, Related AEs and AEs leading to Discontinuation in phase 2a subjects.
Time Frame: 12 months
Population: The safety population (all patients) were analyzed for dose limiting toxicities and treatment emergent adverse events. Treatment totals include all patients that received the specific dose at any point during the study.
Measure: Number; unit: Patients with event
Arm/Group | Phase 2a Expansion Cohort
Number analyzed (Participants) | 5
Patients with event
  At least one TEAE | 5
  At least one Serious TEAE | 2
  At least one severe TEAE | 5
  At least one related TEAE | 5
  At least one TEAE leading to discontinuation | 2

3. Secondary Outcome: Evaluate the Pharmacokinetic (PK) Profile of CRLX301
Description: Area under the concentration vs time curve of released docetaxel in blood and/or urine specimens of patients receiving at least 1 dose of CRLX301.
Time Frame: 2.5 years
Measure: Mean (Standard Deviation); unit: ng/ml*h
Arm/Group | Schedule 1 Cohort 1 | Schedule 1 Cohort 2 | Schedule 1 Cohort 3 | Schedule 1 Cohort 5 | Schedule 1 Cohort 6 | Schedule 1 Cohort 7 | Schedule 2 Cohort 1 | Schedule 2 Cohort 2 | Schedule 2 Cohort 3 | Schedule 2 Cohort 4
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 6 | 6 | 3 | 4 | 3 | 3
ng/ml*h | 295 (0) | 2197 (0) | 1695 (438) | 3783 (1054) | 3613 (1054) | 4639 (1561) | 1433 (154) | 2205 (731) | 2019 (325) | 2350 (453)

4. Secondary Outcome: Percentage of Participants Stratified by Best Overall Tumor Response
Description: Best overall tumor response will be provided per dose cohort using RECIST 1.1
Time Frame: 2.5 years
Population: All patients treated on study (safety population) were evaluated for overall tumor response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Schedule 1 Cohort 1 | Schedule 1 Cohort 2 | Schedule 1 Cohort 3 | Schedule 1 Cohort 5 | Schedule 1 Cohort 6 | Schedule 1 Cohort 7 | Schedule 2 Cohort 1 | Schedule 2 Cohort 2 | Schedule 2 Cohort 3 | Schedule 2 Cohort 4 | Schedule 2 Cohort 5 | Phase 2a Expansion Cohort
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 6 | 6 | 3 | 4 | 4 | 2 | 4 | 5
percentage of participants
  Complete Response | 0 [0 to 97.5] | 0 [0 to 97.5] | 0 [0 to 70.8] | 0 [0 to 70.8] | 0 [0 to 45.9] | 0 [0 to 45.9] | 0 [0 to 70.8] | 0 [0 to 60.2] | 0 [0 to 60.2] | 0 [0 to 84.2] | 0 [0 to 60.2] | 0 [0 to 52.2]
  Partial Response | 0 [0 to 97.5] | 0 [0 to 97.5] | 0 [0 to 70.8] | 0 [0 to 70.8] | 0 [0 to 45.9] | 0 [0 to 45.9] | 0 [0 to 70.8] | 0 [0 to 60.2] | 25 [0.6 to 80.6] | 0 [0 to 84.2] | 0 [0 to 60.2] | 20 [0.5 to 71.6]
  Stable Disease | 0 [0 to 97.5] | 0 [0 to 97.5] | 66.7 [9.4 to 99.2] | 100 [29.2 to 100] | 16.7 [0.4 to 64.1] | 16.7 [0.4 to 64.1] | 100 [29.2 to 100] | 75 [19.4 to 99.4] | 50 [6.8 to 93.2] | 50 [1.3 to 98.7] | 100 [39.8 to 100] | 40 [5.3 to 85.3]
  Progressive Disease | 100 [2.5 to 100] | 100 [2.5 to 100] | 33.3 [0.8 to 90.6] | 0 [0 to 70.8] | 66.7 [22.3 to 95.7] | 16.7 [0.4 to 64.1] | 0 [0 to 70.8] | 25 [0.6 to 80.6] | 25 [0.6 to 80.6] | 50 [1.3 to 98.7] | 0 [0 to 60.2] | 20 [0.5 to 71.6]
  Not Evaluated | 0 [0.0 to 97.5] | 0 [0 to 97.5] | 0 [0 to 70.8] | 0 [0 to 70.8] | 0 [0 to 45.9] | 0 [0 to 45.9] | 0 [0 to 70.8] | 0 [0 to 60.2] | 0 [0 to 60.2] | 0 [0 to 84.2] | 0 [0 to 60.2] | 0 [0 to 52.2]

ADVERSE EVENTS:
Time Frame: All AEs were collected occurring during the study period from the time of the first dose to the last day of the 30-day post-treatment follow-up period.
Arm/Group | Schedule 1 Cohort 1 | Schedule 1 Cohort 2 | Schedule 1 Cohort 3 | Schedule 1 Cohort 5 | Schedule 1 Cohort 6 | Schedule 1 Cohort 7 | Schedule 2 Cohort 1 | Schedule 2 Cohort 2 | Schedule 2 Cohort 3 | Schedule 2 Cohort 4 | Schedule 2 Cohort 5 | Phase 2a Expansion Cohort
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/1 | 1/3 | 1/3 | 0/6 | 0/6 | 0/3 | 2/4 | 0/4 | 0/2 | 0/4 | 1/5
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 3/3 | 3/3 | 1/6 | 3/6 | 1/3 | 2/4 | 1/4 | 1/2 | 0/4 | 2/5
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 3/3 | 3/3 | 6/6 | 6/6 | 3/3 | 4/4 | 4/4 | 2/2 | 4/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Schedule 1 Cohort 1 (N=1) | Schedule 1 Cohort 2 (N=1) | Schedule 1 Cohort 3 (N=3) | Schedule 1 Cohort 5 (N=3) | Schedule 1 Cohort 6 (N=6) | Schedule 1 Cohort 7 (N=6) | Schedule 2 Cohort 1 (N=3) | Schedule 2 Cohort 2 (N=4) | Schedule 2 Cohort 3 (N=4) | Schedule 2 Cohort 4 (N=2) | Schedule 2 Cohort 5 (N=4) | Phase 2a Expansion Cohort (N=5)
Injection site infection (Infections and infestations) | NA | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0)
Oesohageal stenosis (Gastrointestinal disorders) | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0)
Pain (General disorders) | NA | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0)
Pyrexia (General disorders) | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0)
Fall (Injury, poisoning and procedural complications) | NA | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | NA | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | 1 (1)
Liver function test abnormal (Investigations) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | NA | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | NA | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0)
Anaemia (Blood and lymphatic system disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | 0 (0)
Atrial fibrillation (Cardiac disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | 0 (0)
Asthenia (General disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | 0 (0)
Urinary tract infection (Infections and infestations) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 1 (2)
Haematuria (Renal and urinary disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Schedule 1 Cohort 1 (N=1) | Schedule 1 Cohort 2 (N=1) | Schedule 1 Cohort 3 (N=3) | Schedule 1 Cohort 5 (N=3) | Schedule 1 Cohort 6 (N=6) | Schedule 1 Cohort 7 (N=6) | Schedule 2 Cohort 1 (N=3) | Schedule 2 Cohort 2 (N=4) | Schedule 2 Cohort 3 (N=4) | Schedule 2 Cohort 4 (N=2) | Schedule 2 Cohort 5 (N=4) | Phase 2a Expansion Cohort (N=5)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (5) | 2 (3) | 2 (2) | 1 (4) | 2 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 3 (12) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 5 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Episcleritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (4) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distention (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 3 (3) | 1 (1) | 2 (2) | 1 (2) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 2 (3) | 1 (1) | 1 (4) | 2 (2) | 2 (3) | 2 (5) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 2 (3) | 3 (3) | 3 (3) | 0 (0) | 2 (3) | 2 (4) | 2 (6) | 1 (1) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (2) | 2 (2) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 3 (5) | 2 (2) | 3 (7) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (3) | 3 (8) | 5 (6) | 4 (9) | 2 (3) | 3 (5) | 4 (10) | 2 (5) | 4 (10) | 3 (4)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
candida infection (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 1 (3)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 2 (3) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 4 (5) | 2 (3) | 2 (4) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood cholesterol incrased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Electrocardiogram (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (5) | 0 (0)
Reticulocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Waist circumference increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 2 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 5 (7) | 1 (1) | 1 (1) | 4 (9) | 2 (6) | 2 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (3) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 2 (6) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (9) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 2 (3) | 4 (4) | 1 (1) | 1 (1) | 4 (7) | 2 (3) | 3 (4) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 2 (3) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 2 (3) | 0 (0) | 2 (3) | 3 (8) | 1 (2) | 2 (5) | 2 (5)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 0 (0) | 3 (7) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 1 (2) | 1 (2) | 2 (3) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 2 (4) | 1 (5) | 1 (2) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Nail bed tenderness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmenation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (6) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-12-16): https://cdn.clinicaltrials.gov/large-docs/77/NCT02380677/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT02380677/SAP_001.pdf